CLINICAL TRIAL: NCT03939572
Title: Harnessing Mindset in 21st Century Healthcare: Leveraging Mindset in Health Technology
Brief Title: Effects of Physical Activity Adequacy Mindsets on Health and Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Alia Crum, Assistant Professor of Psychology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 36098; DP2AT009511 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-05-07 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Activity Adequacy Mindsets
Keywords: Psychological mindsets; Physical activity; Wearable fitness trackers
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Accurate step count feedback (Active Comparator): All arms are given identical instructions in the onboarding session, including information about the study purpose and Apple Watch. They complete the same set of physiological, cognitive, and psychological measures and receive an Apple Watch to wear for the following 5 weeks. Throughout the 5 weeks, participants complete short daily surveys and longer weekly surveys. Finally, participants come in for an "offboarding" lab session in which the same measures are collected as in the onboarding session.
  In this arm, participants' Apple Watches will simply display their accurate step count.
  Interventions: Behavioral: Accurate step count feedback
- Deflated step count feedback (Experimental): All arms are given identical instructions in the onboarding session, including information about the study purpose and Apple Watch. They complete the same set of physiological, cognitive, and psychological measures and receive an Apple Watch to wear for the following 5 weeks. Throughout the 5 weeks, participants complete short daily surveys and longer weekly surveys. Finally, participants come in for an "offboarding" lab session in which the same measures are collected as in the onboarding session.
  In this arm, participants' Apple Watches will display a deflated step count.
  Interventions: Behavioral: Deflated step count feedback
- Inflated step count feedback (Experimental): All arms are given identical instructions in the onboarding session, including information about the study purpose and Apple Watch. They complete the same set of physiological, cognitive, and psychological measures and receive an Apple Watch to wear for the following 5 weeks. Throughout the 5 weeks, participants complete short daily surveys and longer weekly surveys. Finally, participants come in for an "offboarding" lab session in which the same measures are collected as in the onboarding session.
  In this arm, participants' Apple Watches will display an inflated step count.
  Interventions: Behavioral: Inflated step count feedback
- Accurate feedback + mindset intervention (Experimental): All arms are given identical instructions in the onboarding session, including information about the study purpose and Apple Watch. They complete the same set of physiological, cognitive, and psychological measures and receive an Apple Watch to wear for the following 5 weeks. Throughout the 5 weeks, participants complete short daily surveys and longer weekly surveys. Finally, participants come in for an "offboarding" lab session in which the same measures are collected as in the onboarding session.
  In this arm, participants' Apple Watches will display their accurate step count. Additionally, participants in this arm will receive a meta-mindset intervention.
  Interventions: Behavioral: Accurate feedback + mindset intervention

INTERVENTIONS:
Behavioral: Accurate step count feedback — After one week of baseline step count measurement, participants will receive the intervention. Starting day 8, participants' Apple Watches will start displaying their step count. In this arm, they will simply see their accurate step count.
  Arms: Accurate step count feedback
Behavioral: Deflated step count feedback — After one week of baseline step count measurement, participants will receive the intervention. Starting day 8, participants' Apple Watches will start displaying their step count. In this arm, they will see their step count deflated by 40% (i.e., their step count multiplied by 0.6).
  Arms: Deflated step count feedback
Behavioral: Inflated step count feedback — After one week of baseline step count measurement, participants will receive the intervention. Starting day 8, participants' Apple Watches will start displaying their step count. In this arm, they will see their step count inflated by 40% (i.e., their step count multiplied by 1.4).
  Arms: Inflated step count feedback
Behavioral: Accurate feedback + mindset intervention — After one week of baseline step count measurement, participants will receive the intervention. Starting day 8, participants' Apple Watches will start displaying their step count. In this arm, they will simply see their accurate step count.
  Additionally, participants in this arm will receive a meta-mindset intervention in the first weekly survey on day 7, which consists of a series of videos and reflection exercises to teach participants about the power of mindsets and encourage them to choose adaptive mindsets that will benefit their health. There are also short booster reflection exercises in all subsequent daily and weekly surveys, reinforcing the message about adaptive mindsets.
  Arms: Accurate feedback + mindset intervention

SUMMARY:
It is widely known that physical activity is important for health and wellbeing, yet most Americans do not meet recommended levels of activity. People may commonly believe that only the actual amount of physical activity matters for health and wellbeing. However, the investigators propose that individuals' mindsets about the adequacy of their level of physical activity and its corresponding health consequences (activity adequacy mindsets) affect health outcomes, over and above their actual level of physical activity. In recent years, health technologies such as wearable fitness trackers have become popular tools to promote higher levels of physical activity. This study leverages the tracking and feedback capabilities of Apple Watch to study the effects of mindsets about physical activity on health and wellbeing, as well as the pathways through which these effects may occur.

DETAILED DESCRIPTION:
Study Overview: This study examines how individuals' mindsets about the adequacy of their level of physical activity and its corresponding health consequences (activity adequacy mindsets) affect health outcomes. Participants attend an "onboarding" lab session in which they complete physiological, cognitive, and psychological measures and receive an Apple Watch to wear for the following 5 weeks. The Watch is equipped with a step count tracking app. No step count feedback is provided in week 1 as a baseline; starting in week 2, participants are randomized to 4 conditions in which either 1) accurate, 2) inflated, or 3) deflated step count is displayed on the watch in order to manipulate participants' perceived physical activity, independently of their actual physical activity. In condition 4, participants receive a meta-mindset intervention in addition to accurate step count feedback. Throughout the 5 weeks, participants complete short daily surveys and longer weekly surveys administered online. Finally, participants come in for an "offboarding" lab session in which the same measures are collected as in the onboarding session.

Participants: Participants will be 160 healthy adults recruited from the community, 40 per condition.

Main Hypotheses: This is a largely exploratory study, examining various mechanisms through which activity adequacy mindsets may affect health and wellbeing. Tests include (but are not limited to) the following key hypotheses:

H1) Inflated step count feedback (compared to accurate feedback) leads to a more positive activity adequacy mindset, and deflated feedback (compared to accurate feedback) leads to a more negative activity adequacy mindset (see Primary Outcome Measures).

H2) Activity adequacy mindset influences health and wellbeing (see Primary Outcome Measures) over and above actual physical activity.

H3) Activity adequacy mindset influences health and wellbeing through various mechanisms (see Secondary Outcome Measures):

H3a) Affective mechanism: A more positive (vs. negative) activity adequacy mindset leads to more positive everyday affect (incl. higher satisfaction, lower anxiety, lower stress). Positive affect in turn improves health and wellbeing.

H3b) Motivational/ behavioral mechanism: A more positive (vs. negative) activity adequacy mindset leads to higher motivation to exercise and improve one's health, as well as higher exercise self-efficacy. Higher motivation and self-efficacy in turn lead to higher levels of actual physical activity, which in turn improve health and wellbeing.

H3c) Placebo mechanism: A more positive (vs. negative) activity adequacy mindset directly improves health and wellbeing through placebo/ nocebo effects.

H4) A meta-mindset intervention teaching people about activity adequacy mindsets leads them to adopt more positive mindsets, which in turn predicts improved health and wellbeing through the mechanisms described under H3. That is, compared to accurate step count feedback only, accurate feedback plus meta-mindset intervention leads to improved health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Low level of physical activity in the prior six months, as indicated by self-report
* Walking as primary source of physical activity in the prior six months, as indicated by self-report
* Ability to understand study procedures and to comply with them for the entire length of the study.

Exclusion Criteria:

* Candidates who answer affirmatively to any of the Physical Activity Readiness Questionnaire (PAR-Q) items will be excluded, unless they get clearance from a physician that they are able to participate in the study.
* Candidates who report pregnancy will be excluded, as natural changes in weight and body composition during pregnancy would invalidate our results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Perceived Amount of Exercise Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in daily and weekly surveys, and at end of study (offboarding session)
  Perceived Amount of Exercise (manipulation check), measured via 1-item self-report in all surveys. The full item is "Overall, how much exercise did you get today?", range 1 (None at all) - 5 (A great deal), with high values considered a better outcome.
Change in Activity Adequacy Mindset Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in weekly surveys, and at end of study (offboarding session)
  Activity Adequacy Mindset (key mediator) measured via self-report in onboarding/ offboarding surveys (7 items) and weekly surveys (shortened, 5 items). This scale ranges from 1 - 7, with higher values representing better outcomes. The items will be combined in a composite score by averaging.
Change in Physical Health Over 5 Weeks | 5 weeks: measured at baseline (onboarding session) and end of study (offboarding session); except average daily heart rate, which is based on Apple Watch HR recordings measured approx. every 20 minutes when participant is wearing watch during the 5 weeks
  Physical Health measures are BMI (calculated from self-reported height and weight measured in lab, BMI = kg/m^2); Body fat percentage (measured on lab scale); Resting systolic and diastolic blood pressure (measured in lab); Resting heart rate (HR) (measured in lab); Average daily heart rate (measured by Apple Watch heart rate sensor); VO2max, approximated through the Canadian Home Fitness Test (based on post-exercise HR measured in lab); Perceived general health (measured via 1-item self-report); Perceived fitness (measured via 1-item self-report); Physical function and pain (measured via PROMIS-29 Profile v2.0 questionnaire). All measures will be factor analyzed and combined into a summary score (average of standardized scores weighted by variables' factor loading), provided factor analysis shows that they load onto one factor (i.e., rotated factor loadings of >= |0.4|). Measures will also be analyzed separately for exploratory purposes.
Change in Mental Health Over 5 Weeks | 5 weeks: measured at baseline (onboarding session) and end of study (offboarding session)
  Anxiety, depressive symptoms, ability to participate in social roles and activities, sleep disturbance, fatigue (measured via PROMIS (Patient-Reported Outcomes Measurement Information System)-29 Profile v2.0 questionnaire), and stress (measured via Perceived Stress Scale, PSS). Each PROMIS subscale ranges from 1-5, with higher values representing better outcomes. Items will be averaged into subscale composite scores. The PSS ranges from 1-5, with higher values representing worse outcomes. PSS items will be averaged into a composite score. All measures will be factor analyzed and combined into a summary score (average of standardized scores weighted by variables' factor loading), provided factor analysis shows that they load onto one factor (i.e., rotated factor loadings of >= |0.4|). Measures will also be analyzed separately for exploratory purposes.
Change in Cognitive Function Over 5 Weeks | 5 weeks: measured at baseline (onboarding session) and end of study (offboarding session)
  Stroop task performance

SECONDARY OUTCOMES:
Change in Affect Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in daily and weekly surveys, and at end of study (offboarding session)
  Measured via self-report (Affect Valuation Index, AVI, and 2 items measuring stress/ anxiety). AVI items range from 1-5, with higher scores indicating higher frequency of any given emotion. Items will be averaged into 8 subscale composite scores according to the AVI protocol by averaging. Items measuring stress/ anxiety range from 1-5 with higher scores representing worse outcomes. All measures will be factor analyzed and combined into a summary score (average of standardized scores weighted by variables' factor loading), provided factor analysis shows that they load onto one factor (i.e., rotated factor loadings of >= |0.4|). Measures will also be analyzed separately for exploratory purposes.
Change in Self-Efficacy for Exercise Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in weekly surveys, and at end of study (offboarding session)
  Measured via self-report (Self-Efficacy for Exercise scale). Items range from 1-5, with higher values representing better outcomes. Items will be averaged into a composite scale.
Change in Motivation for exercise and health promotion Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in weekly surveys, and at end of study (offboarding session)
  Measured via self-report (2 items measuring exercise motivation and health promotion motivation). Items range from 1-5, with higher values representing better outcomes. Items will be averaged into a composite scale.
Change in Physical Activity Behavior Over 5 Weeks | 5 weeks: Step count measured by Apple Watch every ~ 15 min when participant is wearing watch during the 5 weeks; IPAQ and custom physical activity measure assessed in onboarding/ offboarding sessions, and the latter also in weekly surveys
  Physical activity is measured via daily step count tracked by Apple Watch, and via self-report (IPAQ, and a measure adapted from NHANES for this study). All measures will be factor analyzed and combined into a summary score (average of standardized scores weighted by variables' factor loading), provided factor analysis shows that they load onto one factor (i.e., rotated factor loadings of >= |0.4|). Measures will also be analyzed separately for exploratory purposes.
Change in Other Health Behaviors (diet, sleep, drinking, smoking) Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in weekly surveys, and at end of study (offboarding session)
  Measured via self-report (9 items). All measures will be factor analyzed and combined into a summary score (average of standardized scores weighted by variables' factor loading), provided factor analysis shows that they load onto one factor (i.e., rotated factor loadings of >= |0.4|). Measures will also be analyzed separately for exploratory purposes.
Change in Process Mindset Over 5 Weeks | 5 weeks: measured at baseline (onboarding session), in one of the weekly surveys, and at end of study (offboarding session)
  Exercise process mindset and Health process mindset are measured via self-report (7 items per scale). Items range from 1-4, with higher values representing better outcomes. Items will be averaged into two composite scores (General Process Mindset and Exercise Process Mindset). If items from both subscales have sufficient reliability (Cronbach's alpha > 0.7), they will be averaged into one composite scale.

CONTACTS AND LOCATIONS:
Overall Officials: Alia J Crum, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
If made publicly available, all data will be de-identified and the anonymous data will be shared with researchers on the Open Science Framework

REFERENCES:
- [Derived] Zahrt OH, Evans K, Murnane E, Santoro E, Baiocchi M, Landay J, Delp S, Crum A. Effects of Wearable Fitness Trackers and Activity Adequacy Mindsets on Affect, Behavior, and Health: Longitudinal Randomized Controlled Trial. J Med Internet Res. 2023 Jan 25;25:e40529. doi: 10.2196/40529. PMID 36696172